CLINICAL TRIAL: NCT01301378
Title: Comparison of Porcine Submucosal Tissue Patch Graft (KeraSys) Versus Processed Pericardium Patch Graft (Tutoplast) in Glaucoma Drainage Implant Surgery Using a Molteno 3 Shunt
Brief Title: Patch Graft Material Safety and Effectiveness in Covering Glaucoma Drainage Device Tube
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: kerasys had more erosions than tutoplast
Sponsor: Wills Eye (Other)
Collaborators: IOP Ophthalmics (Unknown)
Responsible Party: Principal Investigator, Marlene Moster, MD, Marlene Moster, MD Principal Investigator, Wills Eye Institute Glaucoma Department, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-956 KeraSys
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Primary Open Angle Glaucoma; Primary Angle Closure Glaucoma; Pseudoexfoliation Glaucoma; Pigmentary Glaucoma; Traumatic Glaucoma; Uveitic Glaucoma; Neovascular Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma, Angle-Closure; Exfoliation Syndrome; Glaucoma, Neovascular | interventions — Tutoplast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KeraSys Tissue Patch Graft (Active Comparator): 20 patients needing a Molteno 3 glaucoma drainage shunt implant will receive the KeraSys patch graft
  Interventions: Procedure: Molteno 3 glaucoma drainage shunt
- Tutoplast tissue patch graft (Active Comparator): 20 patients need Molteno 3 glaucoma drainage surgery will receive tutoplast patch graft
  Interventions: Procedure: Molteno 3 glaucoma drainage shunt

INTERVENTIONS:
Procedure: Molteno 3 glaucoma drainage shunt — Patients needing glaucoma drainage surgery
  Other Names: Porcine Submucosal Tissue Patch Graft (Kerasys); Processed Pericardium Patch Graft (Tutoplast)

SUMMARY:
The investigators hypothesize that KeraSys is a safe as Tutoplast to cover the tube of the Molteno 3 glaucoma drainage device during surgery

DETAILED DESCRIPTION:
This study compares patients who will undergo Molteno 3 shunt implant surgery with 1 group receiving KeraSys patch graft and the 2nd group receiving Tutoplast patch graft. The investigators will examine the efficacy and safety of KeraSys in comparison with Tutoplast and monitor the long term effectiveness for preventing tube erosion in Molteno 3 tube shunt surgery for 1 year.

ELIGIBILITY:
Inclusion Criteria:

Patients with primary open-glaucoma (POAG), primary angle-closure glaucoma (PACG), pseudoexfoliation, pigmentary, traumatic, uveitic or neovascular glaucoma

Exclusion Criteria:

1. Age ≤ 18 years old.
2. Any type of glaucoma other than those listed in the inclusion criteria.
3. Less than 3 months of other ocular surgery.
4. Active thyroid-related immune orbitopathy, carotid-cavernous fistula, Sturge Weber syndrome, orbital tumors or orbital congestive disease.
5. Patients with connective tissue disorder.
6. Patients with congenital or developmental glaucoma.
7. Patients with severe dry eye syndrome.
8. Patients with any surgical procedure involving revision, removal, or change of the existing glaucoma tube shunt.
9. Patients undergoing any surgical concomitant surgical procedure involving the posterior segment.
10. Patients with active scleritis, history of ocular trauma including chemical burn, chronic ocular inflammatory disease, or ocular surface disease.
11. Patients with any prior history of allergy to the active compound.
12. Pregnancy or breast-feeding.
13. Patients enrolled in other prospective clinical trials.
14. Patients that plan to use contact lens after surgery.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Kerasys safety | one day, week one, 1 month, 3 month, 6 month, and 1 year
  The patch graft will be graded on appearance at each visit by slit lamp for tube erosion and conjunctival retraction.

SECONDARY OUTCOMES:
Long term efficacy of Kerasys and Tutoplast in Molteno 3 glaucoma shunt surgery | 1 month, 3 month, 6 month, 1 year
  The thickness of the patch graft will be measured by anterior segment OCT and anterior segment photos.

CONTACTS AND LOCATIONS:
Overall Officials: Marlene M Moster, MD, Principal Investigator — Wills Eye Institute Glaucoma Department
Locations (1):
- Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lankaranian D, Reis R, Henderer JD, Choe S, Moster MR. Comparison of single thickness and double thickness processed pericardium patch graft in glaucoma drainage device surgery: a single surgeon comparison of outcome. J Glaucoma. 2008 Jan-Feb;17(1):48-51. doi: 10.1097/IJG.0b013e318133fc49. PMID 18303385